CLINICAL TRIAL: NCT02475837
Title: A Double-blind, Randomized, Placebo Controlled Pilot Trial to Evaluate the Safety and Efficacy of Vorapaxar in Maturation of Arteriovenous Fistulae for Hemodialysis Access
Brief Title: Vorapaxar Study for Maturation of AV Fistulae for Hemodialysis Access
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ken Mahaffey (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Ken Mahaffey, Co Investigator, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 33763
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: AV Fistula
MeSH Terms: conditions — Arteriovenous Fistula | interventions — vorapaxar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Vorapaxar intervention (Active Comparator): This arm will receive the study drug: Vorapaxar sulfate.
  The investigators expect to enroll 128 patients. Patients will be assigned to treatment groups with a 1:1 randomization in blocks of 4 at the conclusion of the AV fistula creation. Patients will be stratified based on fistula location (lower arm versus upper arm).
  Interventions: Drug: Vorapaxar sulfate
- Placebo intervention (Placebo Comparator): This arm will receive the matching placebo.
  The investigators expect to enroll 128 patients. Patients will be assigned to treatment groups with a 1:1 randomization in blocks of 4 at the conclusion of the AV fistula creation. Patients will be stratified based on fistula location (lower arm versus upper arm).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vorapaxar sulfate — The study drug (12-week supply of study drug) will be dispensed to enrolled patients on the first day following surgery.
  Other Names: Zontivity
  Arms: Vorapaxar intervention
Drug: Placebo — The placebo will match the study drug, vorapaxar sulfate, in appearance. A 12-week supply will be dispensed to enrolled patients on the first day following surgery.
  Arms: Placebo intervention

SUMMARY:
The Objectives of this study are:

1. To determine if vorapaxar safely improves arteriovenous (AV) fistula functional maturation when administered during the maturation process compared with placebo.
2. To determine if vorapaxar safely improves AV fistula patency, allowing for secondary procedures to aid in fistula maturation compared with placebo.
3. To determine if vorapaxar safely facilitates successful cannulation of AV fistulas for hemodialysis compared with placebo.

This is a randomized placebo-controlled double-blind pilot trial. Study procedures will be conducted at Stanford University Medical Center, and standard-of-care (SOC) procedures will be conducted at Stanford and it's affiliated hospitals (Veteran's Affairs Palo Alto Health Care System and the Stanford Vascular Surgery Clinic at Valley Medical Center). The investigators expect to enroll 128 patients. Patients will be assigned to treatment groups with a 1:1 randomization in blocks of 4 at the conclusion of the AV fistula creation. Patients will be stratified based on fistula location (lower arm versus upper arm).

DETAILED DESCRIPTION:
Objectives:

1. To determine if vorapaxar safely improves arteriovenous (AV) fistula functional maturation when administered during the maturation process compared with placebo.
2. To determine if vorapaxar safely improves AV fistula patency, allowing for secondary procedures to aid in fistula maturation compared with placebo.
3. To determine if vorapaxar safely facilitates successful cannulation of AV fistulas for hemodialysis compared with placebo.

This is a randomized placebo-controlled double-blind pilot trial. Study procedures will be conducted at Stanford University Medical Center, and standard-of-care (SOC) procedures will be conducted at Stanford and it's affiliated hospitals (Veteran's Affairs Palo Alto Health Care System and the Stanford Vascular Surgery Clinic at Valley Medical Center). The investigators expect to enroll 128 patients. Patients will be assigned to treatment groups with a 1:1 randomization in blocks of 4 at the conclusion of the AV fistula creation. Patients will be stratified based on fistula location (lower arm versus upper arm).

Participation in this study will not affect standard care of patients with AV fistulae receiving hemodialysis. The only additional treatment is administration of the study drug or placebo and additional monitoring, including one additional ultrasound, for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Receiving or planning to receive maintenance hemodialysis
3. Ability to sign informed consent
4. 3 mm venous diameter within recipient vein

Exclusion Criteria:

1. History of stroke, transient ischemic attack or intracranial hemorrhage
2. History of or high level of suspicion for, severe arterial insufficiency of the hand
3. Indication or ongoing therapy with other antiplatelet agents, other than aspirin 81 mg daily
4. Indication or ongoing therapy with anticoagulants, including warfarin, low molecular weight heparin, factor Xa inhibitors or direct thrombin and other inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Mell, MD, MS, Principal Investigator — Stanford University; Kenneth W Mahaffey, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Univeristy, Stanford, California, United States

REFERENCES:
- [Background] Brescia MJ, Cimino JE, Appel K, Hurwich BJ. Chronic hemodialysis using venipuncture and a surgically created arteriovenous fistula. N Engl J Med. 1966 Nov 17;275(20):1089-92. doi: 10.1056/NEJM196611172752002. No abstract available. PMID 5923023
- [Background] Andrassy K, Malluche H, Bornefeld H, Comberg M, Ritz E, Jesdinsky H, Mohring K. Prevention of p.o. clotting of av. cimino fistulae with acetylsalicyl acid. Results of a prospective double blind study. Klin Wochenschr. 1974 Apr 1;52(7):348-9. doi: 10.1007/BF01468835. No abstract available. PMID 4600820
- [Background] Crowther MA, Clase CM, Margetts PJ, Julian J, Lambert K, Sneath D, Nagai R, Wilson S, Ingram AJ. Low-intensity warfarin is ineffective for the prevention of PTFE graft failure in patients on hemodialysis: a randomized controlled trial. J Am Soc Nephrol. 2002 Sep;13(9):2331-7. doi: 10.1097/01.asn.0000027356.16598.99. PMID 12191977
- [Background] Fiskerstrand CE, Thompson IW, Burnet ME, Williams P, Anderton JL. Double-blind randomized trial of the effect of ticlopidine in arteriovenous fistulas for hemodialysis. Artif Organs. 1985 Feb;9(1):61-3. doi: 10.1111/j.1525-1594.1985.tb04349.x. PMID 3888153
- [Background] Osborn G, Escofet X, Da Silva A. Medical adjuvant treatment to increase patency of arteriovenous fistulae and grafts. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD002786. doi: 10.1002/14651858.CD002786.pub2. PMID 18843633
- [Background] Kaufman JS. Antithrombotic agents and the prevention of access thrombosis. Semin Dial. 2000 Jan-Feb;13(1):40-6. doi: 10.1046/j.1525-139x.2000.00012.x. No abstract available. PMID 10740671
- [Background] Dember LM, Kaufman JS, Beck GJ, Dixon BS, Gassman JJ, Greene T, Himmelfarb J, Hunsicker LG, Kusek JW, Lawson JH, Middleton JP, Radeva M, Schwab SJ, Whiting JF, Feldman HI; DAC Study Group. Design of the Dialysis Access Consortium (DAC) Clopidogrel Prevention of Early AV Fistula Thrombosis Trial. Clin Trials. 2005;2(5):413-22. doi: 10.1191/1740774505cn118oa. PMID 16317810
- [Background] Hirano K. The roles of proteinase-activated receptors in the vascular physiology and pathophysiology. Arterioscler Thromb Vasc Biol. 2007 Jan;27(1):27-36. doi: 10.1161/01.ATV.0000251995.73307.2d. Epub 2006 Nov 9. PMID 17095716
- [Background] Morrow DA, Braunwald E, Bonaca MP, Ameriso SF, Dalby AJ, Fish MP, Fox KA, Lipka LJ, Liu X, Nicolau JC, Ophuis AJ, Paolasso E, Scirica BM, Spinar J, Theroux P, Wiviott SD, Strony J, Murphy SA; TRA 2P-TIMI 50 Steering Committee and Investigators. Vorapaxar in the secondary prevention of atherothrombotic events. N Engl J Med. 2012 Apr 12;366(15):1404-13. doi: 10.1056/NEJMoa1200933. Epub 2012 Mar 24. PMID 22443427
- [Background] Tricoci P, Huang Z, Held C, Moliterno DJ, Armstrong PW, Van de Werf F, White HD, Aylward PE, Wallentin L, Chen E, Lokhnygina Y, Pei J, Leonardi S, Rorick TL, Kilian AM, Jennings LH, Ambrosio G, Bode C, Cequier A, Cornel JH, Diaz R, Erkan A, Huber K, Hudson MP, Jiang L, Jukema JW, Lewis BS, Lincoff AM, Montalescot G, Nicolau JC, Ogawa H, Pfisterer M, Prieto JC, Ruzyllo W, Sinnaeve PR, Storey RF, Valgimigli M, Whellan DJ, Widimsky P, Strony J, Harrington RA, Mahaffey KW; TRACER Investigators. Thrombin-receptor antagonist vorapaxar in acute coronary syndromes. N Engl J Med. 2012 Jan 5;366(1):20-33. doi: 10.1056/NEJMoa1109719. Epub 2011 Nov 13. PMID 22077816
- [Background] Kosoglou T, Kraft WK, Kumar B, Statkevich P, Xuan F, Ma L, Jennings LK, Schiller JE, Langdon RB, Cutler DL. Pharmacokinetics and pharmacodynamics of the novel PAR-1 antagonist vorapaxar in patients with end-stage renal disease. Eur J Clin Pharmacol. 2012 Jul;68(7):1049-56. doi: 10.1007/s00228-012-1217-6. Epub 2012 Feb 8. PMID 22315147

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants were enrolled, 13 were randomized.
Groups:
- Vorapaxar Intervention: Participants were randomized to receive vorapaxar sulfate for 12 weeks (2.5 mg orally once daily).
- Placebo Intervention: Participants were randomized to receive placebo to match vorapaxar sulfate for 12 weeks.
Period: Overall Study
Arm/Group | Vorapaxar Intervention | Placebo Intervention
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorapaxar Intervention | Placebo Intervention | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.0 [45.0 to 66.0] | 62.0 [46.0 to 66.0] | 56.0 [45.0 to 66.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Time to AV Fistula Functional Maturation
Description: Time to AV fistula functional maturation (defined as successful cannulation of the AV fistula for six hemodialysis sessions within three weeks).
Time Frame: up to 238 days
Population: Pre-specified time for assessment of this Outcome Measure was up to 180 days, but data collected is out of window due to delayed and rescheduled visits.
Measure: Median (Inter-Quartile Range); unit: Days to functional maturation
Groups:
- Vorapaxar Intervention: Participants were randomized to receive vorapaxar sulfate for 12 weeks (2.08 mg orally once daily).
Arm/Group | Vorapaxar Intervention | Placebo Intervention
Number analyzed (Participants) | 6 | 7
Days to functional maturation | 169 [96 to 238] | 145 [76 to 197]

2. Secondary Outcome: Count of Participants With AV Fistula Use
Description: Participants able to use their AV fistula for dialysis within 180 days of surgery were considered to have met the outcome.
Time Frame: up to 238 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vorapaxar Intervention | Placebo Intervention
Number analyzed (Participants) | 6 | 7
Participants | 2 | 4

3. Secondary Outcome: Count Participants With AV Fistula Patency
Description: Criteria for outcome: AV fistula patency at 150-180 days, with at least 50% increase in vein diameter by ultrasound compared with preoperative vein diameter measurement.
Time Frame: 150-238 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vorapaxar Intervention | Placebo Intervention
Number analyzed (Participants) | 6 | 7
Participants | 1 | 5

4. Secondary Outcome: Count of All Participants With Bleeding Events
Description: Bleeding events according to GUSTO (criteria for bleeding: Severe, Moderate or Mild) and BARC (bleeding criteria Type 0-5, with 0 being no bleeding and 5 referring to probable or definite fatal bleeding) Criteria
Time Frame: up to 238 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vorapaxar Intervention | Placebo Intervention
Number analyzed (Participants) | 6 | 7
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 238 days
Description: Pre-specified time for assessment of Adverse Events was up to 180 days, but data collected is out of window due to delayed and rescheduled visits.
Arm/Group | Vorapaxar Intervention | Placebo Intervention
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorapaxar Intervention (N=6) | Placebo Intervention (N=7)
Aplastic crisis in setting of sickle cell anemia (Blood and lymphatic system disorders) | 0 | 1
Superior vena cava syndrome (Cardiac disorders) | 1 | 0
Melena due to duodenal ulceration (Gastrointestinal disorders) | 0 | 1
Dilation of left ureteral-ileal stricture (Renal and urinary disorders) | 1 | 0
Shortness of breath due to volume overload (Renal and urinary disorders) | 0 | 1
Renal transplant (Renal and urinary disorders) | 1 | 0
Clogged nephrostomy tube (Renal and urinary disorders) | 1 | 0
Miliary tuberculosis (Infections and infestations) | 0 | 1
Community acquired pneumonia (Infections and infestations) | 0 | 1
Severe fever to due catheter infection (Infections and infestations) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study did not reach its planned enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT02475837/SAP_000.pdf
  • Study Protocol (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT02475837/Prot_001.pdf